CLINICAL TRIAL: NCT04098185
Title: Role of Pleural Fluid Attenuation Value Measurement on Computed Tomography as a Diagnostic Tool for Hemothorax in Traumatic Patients
Brief Title: Role of Pleural Fluid Attenuation Value on CT as a Diagnostic Tool in Traumatic Hemothorax
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Abdelazem Abdelbary, Resident of Diagnostic Radiology, Assiut University
Other Study IDs: CT in traumatic hemothorax
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hemothorax; Traumatic
MeSH Terms: conditions — Hemothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT — Non-contrast Multidetector Computed Tomography will be done for all patients using 16 or 64 MDCT scanner. Standard scanning parameters of chest CT are used with slice thickness 5 mm, 120kv and automated mAs.The evaluation of pleural effusion attenuation will be done using the average measure of 3 slices with greatest amount of fluid. A region of interest (ROI) is placed for measurement of Hounsfield unit values, where pleural fluid is observed to be most intense and the density values of the pleural fluid and of the aorta are quantitatively measured in the same section with taking care not to involve adjacent ribs, lung parenchyma or areas of pleural thickening.

SUMMARY:
To define the potential role of pleural fluid attenuation value determined on computed tomography (CT) for diagnosis of traumatic hemothorax and differentiate it from other pleural effusion.

DETAILED DESCRIPTION:
Hemothorax is defined as blood accumulation in the pleural space. It is a consequence of blunt trauma in 90% of cases. Hemothorax due to blunt trauma mechanisms e.g traffic accidents,sport accidents and falls are among the commonest injuries of the chest. It is manifested in 30-50% of chest trauma cases. In such cases, bleeding might be caused by damage to pulmonary parenchyma or intercostal arteries associated with or without rib fractures and other chest wall tissue injuries including parietal pleura or other thoracic structures. Although other pleural effusion types may also manifest such as chylothorax in case of chest trauma, however fluid detected in pleural space is usually considered blood unless proven not to be. Despite the clinical and radiological findings provide important data about the content of pleural cavity, however tube thoracostomy and diagnostic thoracocentesis are still required to relieve pressure and characterize the fluid. Tube thoracostomy is an invasive procedure which can lead to immediate procedural injuries, infections and pain which can contribute to respiratory failure in patients with chest wall injury. Although needle thoracocentesis is less invasive than tube thoracostomy, however it carries small but definitive risks such as pneumothorax, bleeding and chest wall hematoma. Since hemothorax is a potentially life threatening, it must be diagnosed quickly and accurately and all these unnecessary complications should be avoided. Chest computed tomography [CT] has been accepted as the gold standard imaging study for evaluating chest trauma and usually performed in patients with grossly severe chest trauma, as it helps to detect even small hemothorax.

CT can also allow for more advanced characterization of pleural fluid and distinguish hemothorax from any other types of effusion by means of scaling Hounsfield units as in literature, any attenuation value for pleural fluid between 35 and 70 HU is considered typically blood, so it can be considered as an important non-invasive diagnostic tool for diagnosis of hemothorax in traumatic patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years old
* History of blunt chest trauma
* Having mild to moderate effusion
* CT chest within 1st 24 hours of trauma
* Patients underwent tube thoracostomy or thoracocentesis

Exclusion Criteria:

* Patients in need of emergency transfer to surgery.
* Hemodynamically stable.
* Patients with penetrating trauma.
* Patients with no need for tube thoracostomy or thoracocentesis.
* Patients with minimal effusion.
* Pregnant females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above 18 years old with history of blunt chest trauma and hemodynamically unstable.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Role of pleural fluid attenuation value measurement on CT as a diagnostic tool for traumatic hemothorax | from 1 December 2019 to 1 December 2020
  Measurements of pleural effusion attenuation value on CT to diagnose traumatic hemothorax and differentiate it from other types of pleural effusion.

REFERENCES:
- [Background] Sridhar S, Raptis C, Bhalla S. Imaging of Blunt Thoracic Trauma. Semin Roentgenol. 2016 Jul;51(3):203-14. doi: 10.1053/j.ro.2015.12.002. Epub 2015 Dec 18. No abstract available. PMID 27287951
- [Background] Meyer DM. Hemothorax related to trauma. Thorac Surg Clin. 2007 Feb;17(1):47-55. doi: 10.1016/j.thorsurg.2007.02.006. PMID 17650696
- [Background] Sangster GP, Gonzalez-Beicos A, Carbo AI, Heldmann MG, Ibrahim H, Carrascosa P, Nazar M, D'Agostino HB. Blunt traumatic injuries of the lung parenchyma, pleura, thoracic wall, and intrathoracic airways: multidetector computer tomography imaging findings. Emerg Radiol. 2007 Oct;14(5):297-310. doi: 10.1007/s10140-007-0651-8. Epub 2007 Jul 11. PMID 17623115
- [Background] Miller LA. Chest wall, lung, and pleural space trauma. Radiol Clin North Am. 2006 Mar;44(2):213-24, viii. doi: 10.1016/j.rcl.2005.10.006. PMID 16500204
- [Background] Mirvis SE. Imaging of acute thoracic injury: the advent of MDCT screening. Semin Ultrasound CT MR. 2005 Oct;26(5):305-31. doi: 10.1053/j.sult.2005.08.001. PMID 16274001
- [Background] Hooper C, Lee YC, Maskell N; BTS Pleural Guideline Group. Investigation of a unilateral pleural effusion in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii4-17. doi: 10.1136/thx.2010.136978. No abstract available. PMID 20696692
- [Background] Romero M, Bachler P. Pseudo-hemothorax at computed tomography due to residual contrast media. Clin Imaging. 2014 May-Jun;38(3):333-5. doi: 10.1016/j.clinimag.2014.01.004. Epub 2014 Jan 16. PMID 24559752
- [Background] Kaewlai R, Avery LL, Asrani AV, Novelline RA. Multidetector CT of blunt thoracic trauma. Radiographics. 2008 Oct;28(6):1555-70. doi: 10.1148/rg.286085510. PMID 18936021
- [Background] Gordon CE, Feller-Kopman D, Balk EM, Smetana GW. Pneumothorax following thoracentesis: a systematic review and meta-analysis. Arch Intern Med. 2010 Feb 22;170(4):332-9. doi: 10.1001/archinternmed.2009.548. PMID 20177035
- [Background] Liu F, Huang YC, Ng YB, Liang JH. Differentiatepleural effusion from hemothorax after bluntchest trauma; comparison of computed tomography attenuation values. Journal of AcuteMedicine 2016; 6: 1-6.
- [Background] Cummings KW, Javidan-Nejad C, Bhalla S. Multidetector computed tomography of nonosseous thoracic trauma. Semin Roentgenol. 2014 Apr;49(2):134-42. doi: 10.1053/j.ro.2014.01.002. Epub 2014 Jan 28. No abstract available. PMID 24836489
- [Background] Bolus D, Morgan D, Berland L. Effective use of the Hounsfield unit in the age of variable energy CT. Abdom Radiol (NY). 2017 Mar;42(3):766-771. doi: 10.1007/s00261-017-1052-4. PMID 28132073